CLINICAL TRIAL: NCT02600208
Title: BT13BTθ51 Unrelated and Partially Matched Related Donor Peripheral Stem Cell Transplantation with Alpha Beta T Cell and B Cell Depletion for Patients with Hematologic Malignancies
Brief Title: Peripheral Blood Stem Cell Transplantation for Hematologic Malignancies with Alpha Beta TCell and B Cell Depletion Using the CliniMACS Device
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Julie-An M. Talano (Other)
Collaborators: Miltenyi Biotec, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Julie-An M. Talano, Associate Professor - Department of Pediatrics - Division of Hematology/Oncology, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT13BTθ51
Record Dates: First submitted 2015-10-28; First posted 2015-11-09 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Experimental Arm (Experimental): Alpha Beta T cell depletion is performed for all PBSC grafts using the CliniMACs device
  Interventions: Device: CliniMACs

INTERVENTIONS:
Device: CliniMACs — Depletion of Alpha Beta T cells in the PBSC graft
  Other Names: Alpha/Beta T-Cell Depletion

SUMMARY:
This is a single arm pilot study for patients with hematologic malignancies with alternative donor sources receiving unrelated or partially matched related/Haploidentical mobilized peripheral stem cells (PSCs) using the CliniMACS system for Alpha Beta T cell depletion plus CD19+ B cell depletion to determine efficacy as determined by engraftment and GVHD, and one year leukemia free survival.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate a new method of T cell depletion using the Miltenyi CliniMACS™ device for patients undergoing a peripheral stem cell transplant utilizing either a unrelated donor or partially matched/haploidentical related donor. This new method is called α/β (alpha/beta) T cell depletion and CD19+ B cell depletion. This pilot study will evaluate if this new method of T cell and B cell depletion is a more effective way of removing T cells thus reducing the risk of severe acute and chronic GVHD and result in a durable engraftment.

ELIGIBILITY:
Inclusion Criteria:

Patient:

1. Age. Patient age < 23 years. Both genders and all races eligible.
2. Disease eligibility

Leukemias/lymphomas:

* Acute myeloid leukemia, primary or secondary
* Disease status: remission or <10% bone marrow blasts
* Myelodysplasia
* Acute lymphoblastic leukemia
* Disease status: in hematologic remission
* Chronic myelogenous leukemia:
* Disease status: chronic phase, accelerated phase or blast crisis now in second chronic phase.
* Mixed lineage or biphenotypic acute leukemia
* Lymphoblastic lymphoma
* Disease status: remission
* Burkitt's lymphoma/leukemia:
* Disease status: in remission

Exclusion Criteria:

* Patient

  1. Patients who do not meet disease, organ or infectious criteria.
  2. No suitable donor

Max Age: 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the engraftment of patients receiving unrelated donor or partially matched related donor peripheral stem cells that have T cell depleted and CD19+ B cell depleted using the CliniMACS device. | DAY 42
  Engraftment will be defined using the standard CIBMTR definition of ANC >500 for the first of 3 consecutive days.

SECONDARY OUTCOMES:
Assess the probability of one year leukemia free survival (LFS). | 1 year
  Leukemia relapse is defined as presence of malignant cells in the blood or other body site after initiation of conditioning in a patient previously in remission.
Estimate the incidence and extent of acute and chronic graft vs. host disease. | 1 year
  Acute GVHD will be graded using the standard Glucksberg grading system.
Assess the incidence treatment-related mortality (TRM). | 1 year
  TRM is defined as death from non-disease related causes in the 100 days from stem cell infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Julie-An Talano, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States